CLINICAL TRIAL: NCT00652236
Title: Cost of Long Term Disability in Patients With Chronic Non-Specific Low Back Pain. Three-Year Follow up of a Randomized Trial
Brief Title: Cost of Long Term Disability in Patients With Chronic Non-Specific Low Back Pain
Status: Terminated | Type: Observational
Why Stopped: Study was terminated according the study protocol end of 2007
Sponsor: Klinik Valens (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other); Zurich University of Applied Sciences (Other)
Responsible Party: Bachmann Stefan, MD, Vice Head of Departement of Rheumatology, Rehabilitationszentrum Klinik Valens, CH- 7317 Valens
Other Study IDs: 405340-111500
Record Dates: First submitted 2008-03-27; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Low Back Pain
Keywords: Low back pain; Economics; Cost-effectiveness
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FCT: Patients passing a function- centred rehabilitation
  Interventions: Other: Physiotherapy
- PCT: Patients passing a pain-centred rehabilitation
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The two groups passed an in-patient rehabilitation and a physiotherapy: FCT function-centred vs. PCT pain-centred

SUMMARY:
The purpose of the study was to determine the cost-effectiveness of a function-centred treatment (FCT) compared with a pain-centred treatment (PCT) in patients with chronic low back pain (LBP) in an in-patient setting. Follow-up lasted three years. Direct and indirect costs were recorded by questionnaires sent to health insurances, employers and Swiss Disability Insurance Company.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain, sick leave of 6 weeks during the last 6 months

Exclusion Criteria:

* not able to perform a training program

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Tertiary rehabilitaton centre
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
cost- effectiveness | 3 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bachmann, MD, Principal Investigator — Rehabilitationszentrum Klinik Valens
Locations (1):
- Rehabilitationszentrum Klinik Valens, Valens, Canton of St. Gallen, Switzerland